CLINICAL TRIAL: NCT03605017
Title: The Development of a Virtual Reality Program to Improve Attention in Individuals With TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Krch, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-820-14
Record Dates: First submitted 2018-06-29; First posted 2018-07-30 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: cognitive rehabilitation; attention; executive function
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VREFT: Wonderkin Treatment (Experimental): Administered by computer
  Interventions: Behavioral: Virtual Reality Executive Function Training (VREFT)
- VREFT: Attention Control (Active Comparator): Administered by computer
  Interventions: Behavioral: Virtual Reality Executive Function Training (VREFT)

INTERVENTIONS:
Behavioral: Virtual Reality Executive Function Training (VREFT)

SUMMARY:
The purpose of this research is to investigate the effectiveness of a technique designed to improve divided attention and set-shifting impairments in persons with a traumatic brain injury (TBI). The study is designed to evaluate how well this technique can help people with TBI increase their attention and ability to function better in everyday life.

DETAILED DESCRIPTION:
A pilot study will be conducted to evaluate the effectiveness of a technique designed to improve higher level attention (switching between tasks and multi-tasking) for persons with a traumatic brain injury. 32 individuals with TBI will be recruited. Baseline assessment includes neuropsychological evaluation using traditional measures as well as a completion of a number of questionnaires designed to measure everyday attention and everyday functioning. Participants are random assigned to either the experimental or control groups. Experimental and control treatments include two 60 minute sessions, twice per week, for 5 weeks. Follow-up assessment includes a neuropsychological evaluation using traditional measures as well as a completion of a number of questionnaires designed to measure everyday attention and everyday functioning. Protocol efficacy will be determined by improvements between baseline and follow-up on several objective and functional measures of divided attention and set-shifting.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* diagnosis of TBI
* can read and speak English fluently

Exclusion Criteria:

* prior stroke or neurological disease other than TBI
* unstable or uncontrolled seizures
* currently taking benzodiazepines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-03-26 (Actual); Primary Completion 2022-03-26 (Estimated); Study Completion 2022-03-26 (Estimated)

PRIMARY OUTCOMES:
Total divided attention post-treatment (covarying for baseline performance) | 7 weeks (between pre- and post-testing)
  Comparison between treatment and control groups on post-treatment Auditory Consonant Trigrams
Total set-shifting post-treatment (covarying for baseline performance) | 7 weeks (between pre- and post-testing)
  Comparison between treatment and control groups on post-treatment Stroop interference

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided